CLINICAL TRIAL: NCT03932422
Title: Analysis of Central Hemodynamic Parameters and Sodium Urinary Excretion in Controlled and Resistant Hypertensive Patients
Brief Title: Central Hemodynamic and Sodium Urinary
Acronym: CHASSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Base (Other)
Collaborators: Sao Jose do Rio Preto Medical School (Other)
Responsible Party: Principal Investigator, JOSE FERNANDO VILELA-MARTIN, Principal Investigator and Clinical Professor, Hospital de Base
Other Study IDs: CHASSI
Record Dates: First submitted 2019-04-13; First posted 2019-04-30 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Hypertension
Keywords: hypertension; resistant hypertension; arterial stiffness; sodium urine test
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — The biospecimens retained was urine to analyse the sodium urinary excretion during 24h. Must be done two collects and the data considered it will be the mean between both
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controlled Hypertensive Patients (CHP): Hypertensive patients that have blood pressure less than 140 x 90 mmHg. This parameter must be evaluated by ambulatory blood pressure monitoring
- Resistant Hypertensive Patients (RHP): Hypertensive patients that have blood pressure more than 140 x 90 mmHg and they use three antihypertensive medicines; or hypertensive patients that have blood pressure less than 140 x 90 mmHg, but they use four or more antihypertensive medicines. This parameter must be evaluated by ambulatory blood pressure monitoring.
  Interventions: Diagnostic Test: Evaluate if the individuals are resistant hypertensive patients

INTERVENTIONS:
Diagnostic Test: Evaluate if the individuals are resistant hypertensive patients — Evaluation of the individuals has the objective determine if they are resistant hypertensive patients. This is important because the resistant people have worse prognosis than the controlled people and need more attention from the health professionals. Analysis must be done using the ambulatory blood pressure monitoring.
  Groups: Resistant Hypertensive Patients (RHP)

SUMMARY:
Systemic arterial hypertension is one of major risk factors to development of target organ damage that culminate in cardiovascular diseases such as acute myocardial infarction and stroke. Sodium intake is related with elevation of arterial blood pressure due to rise of cardiac output and of arterial stiffness and it can be estimated by daily sodium excreted in urine 24h. Ambulatory Blood Pressure Monitoring can be used to obtain peripheral and central hemodynamic parameters [arterial stiffness parameters - central blood pressure, pulse wave velocity and augmentation index]. Applanation tonometry also can be used to check same central hemodynamic parameters. Both methods provide us important informations about the patients clinical conditions and help us to infer their prognosis. Therefore, this protocol aims measure the central hemodynamic parameters in hypertensive patients, controlled or resistant, and evaluate their sodium urinary excretion. The hypothesis is the resistant hypertensive patients have parameters higher than controlled hypertensive patients.

DETAILED DESCRIPTION:
The urinary sodium (Na+) will be evaluated by flame photometry. Excretion of urinary sodium will be calculated by multiplying the urinary sodium concentration in mE /L by 24-hour urinary volume. Two to three urinary Na+ samples will be collected within six months.

3.3.3 ABLOOD PRESSURE MONITORING - 24 HOURS Ambulatorial blood pressure monitoring 24-hour will be performed using a Mobil-O-Graph® compact digital device (version 12, ambulatory pressure monitor, 2000, UK). Individuals will be instructed to maintain their normal activities of daily living. The device will be pre-programmed to measure blood pressure within 24 hours at 30-minute intervals every hour during the waking period and at 1-hour intervals during sleep. This device will evaluate the following parameters: systolic and peripheral diastolic blood pressure, mean arterial pressure, pulse pressure, systolic central aortic pressure, central diastolic aortic pressure (cDBP), central pulse pressure (cPP), augmentation index corrected for 75 bpm (AI75%) and pulse wave velocity (PWV).

ELIGIBILITY:
Inclusion Criteria:

* over than 18 years old;
* hypertensive patient for more than four weeks;
* controlled hypertension;
* resistant hypertension;
* regular patient in the local where the study will be done.

Exclusion Criteria:

* chronic renal failure in dyalisis;
* been in the hospital in last 60 days;
* used vasoactive drugs in last 30 days;
* heart failure in III or IV functional class (NYHA);
* pregnant/breastfeeding;
* serious liver disease;
* HIV positive;
* psychiatric diseases that make it difficult to participate;
* stroke or acute myocardial infarction in last 30 days;
* cancer with prognosis less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals will be selected from the hypertensive patients who are assisted in the health service where the study will be performed.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-03-15 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity | The urinary sodium excretion will be evaluated during 24 hours. This evaluation will be done by 2 to 3 times in a period of 6 months. Pulse wave velocity will be also evaluated in this period by the ambulatory blood pressure monitoring 24 hours.
  The investigators has the objective of investigating if the urinary sodium quantity is associated with pulse wave velocity in resistant hypertensive individuals.

CONTACTS AND LOCATIONS:
Overall Officials: José F Vilela-Martin, MD PhD FAHA, Principal Investigator — State Medical School at São José do Rio Preto (FAMERP), São Paulo, Brazil
Locations (1):
- Fundação Faculdade Regional de Medicina (FUNFARME), São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided